CLINICAL TRIAL: NCT00003299
Title: A Randomized Phase III Study Comparing Etoposide and Cisplatin With Etoposide, Cisplatin and Paclitaxel in Patients With Extensive Small Cell Lung Cancer
Brief Title: Cisplatin Plus Etoposide With or Without Paclitaxel in Treating Patients With Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); North Central Cancer Treatment Group (Network); Eastern Cooperative Oncology Group (Network); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-9732; U10CA031946 (NIH); CLB-9732; E-C9732; NCCTG-C9732; SWOG-C9732; CDR0000066238 (Registry Identifier: NCI Physician Desk Reference)
Record Dates: First submitted 1999-11-01; First posted 2004-02-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; Etoposide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cisplatin + Etoposide (Active Comparator)
  Interventions: Drug: cisplatin; Drug: etoposide
- Cisplatin + Etoposide + Paclitaxel (Experimental)
  Interventions: Drug: cisplatin; Drug: etoposide; Drug: paclitaxel

INTERVENTIONS:
Drug: cisplatin
Drug: etoposide
Drug: paclitaxel
  Arms: Cisplatin + Etoposide + Paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known whether cisplatin, etoposide, and paclitaxel are more effective than cisplatin and etoposide alone in treating patients with extensive-stage small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of cisplatin plus etoposide with or without paclitaxel in treating patients with extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether the addition of paclitaxel to standard chemotherapy treatment comprising etoposide and cisplatin improves the survival of patients with extensive stage small cell lung cancer. II. Compare the tumor response rate and failure-free survival of these patients treated with these regimens. III. Describe and compare the toxic effects associated with these regimens in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to performance status and gender. Patients are randomized to one of two treatment arms. Arm I: Patients receive cisplatin IV on day 1 and etoposide IV over 1 hour on days 1-3. Arm II: Patients receive paclitaxel IV over 3 hours on day 1 and cisplatin and etoposide as in arm I. Patients then receive filgrastim (G-CSF) subcutaneously on days 4-18. Treatment repeats in both arms every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients are followed at least every 2 months for 2 years, every 4 months for 1 year, and then at least every 6 months for 2 years.

PROJECTED ACCRUAL: Approximately 670 patients (335 per arm) will be accrued for this study within 16 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically documented extensive stage small cell carcinoma of the bronchus Measurable or evaluable disease No pleural effusions, bone scan abnormalities, or bone marrow biopsies as only evidence of disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: CALGB 0-1 Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL SGOT less than 2 times normal Renal: Serum creatinine no greater than 1.5 mg/dL Cardiovascular: No cardiac disease Pulmonary: No interstitial pneumonia No fibroid lung Other: Not pregnant or nursing Fertile patients must use effective contraception No psychiatric illness No malabsorption disorder No uncontrolled infection No uncontrolled diabetes mellitus No prior or concurrent malignancy within the past 5 years except carcinoma in situ of the cervix or basal cell skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for small cell lung cancer No other concurrent chemotherapy Endocrine therapy: No chronic steroid therapy (except steroids for adrenal failure or hormones for non-disease related conditions) Radiotherapy: No prior pelvic or mediastinal radiotherapy Surgery: Not specified Other: No concurrent anticonvulsants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 587 (Actual)
Dates: Start 1998-04; Primary Completion 2005-06 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
overall survival | Up to 5 years
response rate | Up to 5 years
failure-free survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Harvey B. Niell, MD, Study Chair — Veterans Affairs Medical Center - Memphis; Randolph S. Marks, MD, Study Chair — Mayo Clinic; Alan B. Sandler, MD, Study Chair — Vanderbilt-Ingram Cancer Center; Karen Kelly, MD, Study Chair — University of Colorado, Denver
Locations (20):
- United States (19):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada

REFERENCES:
- [Background] Blackstock AW, Herndon JE 2nd, Paskett ED, Miller AA, Lathan C, Niell HB, Socinski MA, Vokes EE, Green MR; Cancer and Leukemia Group B. Similar outcomes between African American and non-African American patients with extensive-stage small-cell lung carcinoma: report from the Cancer and Leukemia Group B. J Clin Oncol. 2006 Jan 20;24(3):407-12. doi: 10.1200/JCO.2005.02.1436. Epub 2005 Dec 19. PMID 16365181
- [Result] Niell HB, Herndon JE 2nd, Miller AA, Watson DM, Sandler AB, Kelly K, Marks RS, Perry MC, Ansari RH, Otterson G, Ellerton J, Vokes EE, Green MR; Cancer and Leukemia Group. Randomized phase III intergroup trial of etoposide and cisplatin with or without paclitaxel and granulocyte colony-stimulating factor in patients with extensive-stage small-cell lung cancer: Cancer and Leukemia Group B Trial 9732. J Clin Oncol. 2005 Jun 1;23(16):3752-9. doi: 10.1200/JCO.2005.09.071. PMID 15923572
- [Result] Niell HB, Herndon JE, Miller AA, et al.: Randomized phase III intergroup trial (CALGB 9732) of etoposide (VP-16) and cisplatin (DDP) with or without paclitaxel (TAX) and G-CSF in patients with extensive stage small cell lung cancer (ED-SCLC). [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1169, 2002.
- [Derived] Ventz S, Khozin S, Louv B, Sands J, Wen PY, Rahman R, Comment L, Alexander BM, Trippa L. The design and evaluation of hybrid controlled trials that leverage external data and randomization. Nat Commun. 2022 Oct 2;13(1):5783. doi: 10.1038/s41467-022-33192-1. PMID 36184621